CLINICAL TRIAL: NCT04548583
Title: A Phase IB/IIA Study of Remestemcel-L, an Ex-vivo Culture-expanded Adult Allogeneic Bone Marrow Derived Mesenchymal Stem Cell Product for the Treatment of Medically Refractory Crohn's Colitis
Brief Title: Study of Mesenchymal Stem Cells for the Treatment of Medically Refractory Crohn's Colitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Cleveland Clinic (Other)
Collaborators: Mesoblast, Inc. (Industry)
Responsible Party: Principal Investigator, Amy Lightner, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-845
Record Dates: First submitted 2020-09-03; First posted 2020-09-14 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Crohn Colitis
MeSH Terms: conditions — Crohn Disease | interventions — remestemcel-l

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- remestemcel-L (150 million cells) (Experimental): Targeted endoscopic delivery of remestemcel-L, at a dose of 150 million cells into the submucosal layer of the colon wall at baseline
  If at 3 months post injection of remestemcel-L there is clinical, endoscopic or radiographic improvement, patients will receive a second dose of remestemcel-L at a dose of 150 million MSCs (same dose at initial)
  Interventions: Drug: Remestemcel-L
- remestemcel-L (300 million cells) (Experimental): Targeted endoscopic delivery of remestemcel-L, at a dose of 300 million cells into the submucosal layer of the colon wall at baseline.
  If at 3 months post injection of remestemcel-L there is clinical, endoscopic or radiographic improvement, patients will receive a second dose of remestemcel-L at a dose of 300 million MSCs (same dose at initial).
  Interventions: Drug: Remestemcel-L
- Placebo (Placebo Comparator): Direct injection of normal saline into the submucosal layer of the colon wall. If not completely healed after 3 months, participants will then cross over to the treatment group to receive a direct injection of remestemcel-L, at a dose of 150 or 300 million cells into the submucosal layer of the colon wall.
  If at 6 months post injection of remestemcel-L there is clinical, endoscopic or radiographic improvement, patients will receive a second dose of remestemcel-L at a dose of 150 or 300 million MSCs (same dose at initial).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Remestemcel-L — adult allogeneic bone marrow derived mesenchymal stem cell product for the treatment of medically refractory Crohn's colitis
  Arms: remestemcel-L (150 million cells)
Drug: Remestemcel-L — adult allogeneic bone marrow derived mesenchymal stem cell product for the treatment of medically refractory Crohn's colitis
  Arms: remestemcel-L (300 million cells)
Other: Placebo — Normal saline
  Arms: Placebo

SUMMARY:
Crohn's disease has several phenotypes (inflammatory, stricturing, fistulizing) and location (small bowel, ileocecal, colon, and perianal). Approximately one third of patients have inflammation limited to the colon. Up to two thirds will become medically refractory and require a total abdominal colectomy for symptom control. The purpose of this study is to determine the safety and efficacy of using allogeneic bone marrow derived mesenchymal stem cells (MSCs) delivered by targeted endoscopic delivery to treat people for medically refractory Crohn's colitis.

DETAILED DESCRIPTION:
Participants with medically refractory Crohn's colitis will be treated by targeted endoscopic delivery of remestemcel-L, an ex vivo culture expanded allogeneic bone marrow derived mesenchymal stem cell product at a dose of 150 or 300 million. This will be injected into the submucosal layer of the colon and rectal wall.

Patients will receive a second dose of remestemcel-L at a dose of 150 or 300 million MSCs (same dose as initial). If at 3 months post injection of remestemcel-L there is clinical remission, escalation of medical management and/or surgery will be delayed and patients observed. If there is worsening or no improvement in treated patients, then patients will proceed with escalation of medical management or colectomy as per standard of care. Control patients without improvement will cross over to receive remestemcel-L at 3 months and may be retreated at 6 months. All patients will be followed for two years post initial treatment.

There will be a total of 4 cohorts of 3 patients (2 treatment:1 control) receiving the 150 million MSC dose of study drug and a total of 4 cohorts of 3 patients (2 treatment:1 control) receiving 300 million MSCs dose of study drug. This study plans to enroll a total of 24 participants.

The primary endpoint of this study is to determine the safety and feasibility of endoscopic injection of remestemcel-L, an ex vivo culture expanded allogeneic bone marrow derived mesenchymal stem cell product for treatment of medically refractory Crohn's colitis.

ELIGIBILITY:
Inclusion Criteria for all patients to join the protocol

1. Males and Females 18-75 years of age.
2. Crohn's colitis of at least 6 months duration with medically refractory symptoms who has failed one anti-TNF therapy, with a next step of subtotal colectomy or escalation in medical management.
3. Exposure to corticosteroids, 5-ASA drugs, thiopurines, methotrexate, anti-TNF therapy, anti-integrin and anti-interleukin in the past are permitted but a washout period of 4 weeks for any monoclonal antibody is necessary.

   1. If receiving conventional immunomodulators (ie, AZA, 6-MP, or MTX), must have been taking them for ≥12 weeks, and on a stable dose for at least 4 weeks.
   2. If AZA, 6-MP, or MTX has been recently discontinued, it must have been stopped for at least 4 weeks.
   3. If receiving oral 5-ASA compounds, the dose must have been stable for at least 4 weeks.If receiving oral corticosteroids, the dose must be ≤20 mg/day prednisone or its equivalent and must have been stable for at least 4 weeks.
   4. If receiving budesonide, the dose must have been stable for at least 2 weeks.
   5. If oral 5-ASA compounds or oral corticosteroids (including budesonide) have been recently discontinued, they must have been stopped for at least 2 weeks.
4. The following medications/therapies must have been discontinued before first administration of study agent:

   1. TNF-antagonist therapy (eg, infliximab, etanercept, certolizumab, adalimumab, golimumab), vedolizumab, ustekinumab for at least 4 weeks.
   2. Cyclosporine, tacrolimus, or sirolimus, for at least 4 weeks.
   3. 6-thioguanine (6-TG) must have been discontinued for at least 4 weeks.
   4. Rectal corticosteroids (ie, corticosteroids [including budesonide] administered to the
   5. rectum or sigmoid colon via foam or enema or suppository) for at least 2 weeks.
   6. Rectal 5-ASA compounds (ie, 5-ASAs administered to the rectum or sigmoid colon viafoam or enema or suppository) for at least 2 weeks.
   7. Parenteral corticosteroids for at least 2 weeks.
   8. Total parenteral nutrition (TPN) for at least 2 weeks.
   9. Antibiotics for the treatment of UC (eg, ciprofloxacin, metronidazole, or rifaximin) for atleast 2 weeks.
5. No colonic dysplasia and malignancy as ruled out by colonoscopy within 30 days of MSC delivery
6. Ability to comply with protocol
7. Competent and able to provide written informed consent
8. Must have lost response to at least one monoclonal antibody (anti-TNF, anti-interleukin, or anti- integrin therapy), or tofacitinib, or have a contra-indication to biologic therapy

Exclusion Criteria

1. Inability to give informed consent.
2. Clinically significant medical conditions within the six months before administration of MSCs: e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the patient.
3. Specific exclusions;

   1. HIV
   2. Hepatitis B or C
   3. Abnormal AST or ALT at screening defined as > 3x upper limit of normal?
4. History of cancer including melanoma (with the exception of localized skin cancers) within 5 years of study enrollment
5. Investigational drug within one year of study enrollment
6. Pregnant or breast feeding.
7. If patient is of reproductive capacity, unwilling to use adequate birth control measures while they are in the study
8. Fulminant colitis requiring emergency surgery
9. Concurrent active clostridium difficile infection of the colon
10. Concurrent CMV infection of the colon
11. Evidence of colonic perforation
12. Massive hemorrhage from the colon requiring emergent surgery
13. Ulcerative colitis or indeterminate colitis
14. Neoplasia of the colon on preoperative biopsy
15. Presence of an ostomy
16. Three or more prior small bowel resections
17. Colonic stricture that unable to pass an adult colonoscope
18. Active or latent tuberculosis
19. Unable to wean off corticosteroids
20. Patients with primary sclerosing cholangitis
21. Patients with a known allergy to DMSO, porcine and/or bovine proteins. Control patients will have additional criteria that need to be met prior to the patients' crossing over to receive treatment.

Inclusion Criteria for control patients prior to entering the treatment phase:

1. Received placebo at the point of first injection
2. Completed all study visits to date
3. Clinical status has remained the same or improved, not worsened

Exclusion Criteria for control patients who will be entering the treatment phase:

1. Required repeat hospitalization for a colitis flare
2. Given oral and intravenous steroids for a colitis flare
3. Had worsening abdominal pain frequency of bowel movements, blood in stool
4. Desires exclusion from the study to pursue escalation in medical management or surgery
5. Has a colonic perforation that requires surgery
6. Has colonic bleeding that requires surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-11-04 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Treatment related adverse events | Month 3
  The primary endpoint of this study is to determine the safety and feasibility of endoscopic injection of remestemcel-L, an ex vivo expanded allogeneic bone marrow-derived mesenchymal stem cell product, for treatment of medically refractory Crohn's colitis.

SECONDARY OUTCOMES:
Complete clinical healing | Month 3, Month 12
  Number of participants with complete clinical healing post-injection of 150 or 300 million bone marrow allogeneic derived mesenchymal stem cells for the treatment of medically refractory Crohn's colitis.
  Complete healing is defined as: Clinical and endoscopic remission
  Clinical Healing: Normalization of CRP to <2.87 mg per liter, CDAI drops to <150
  Radiographic Healing: MR enterography with improvement of inflammation
  Endoscopic healing: Absence of mucosal ulceration and SES-CD score of 0-5
Clinical response | Month 3, Month 12
  Number of participants with clinical response post-injection of 150 or 300 million allogeneic bone marrow derived mesenchymal stem cell product for the treatment of medically refractory Crohn's colitis.
  Clinical response is defined as:
  Clinical Healing: Normalization of CRP to <2.87 mg per liter, CDAI drops to <150
  Radiographic Healing: MR enterography with improvement of inflammation
  Endoscopic healing: Absence of mucosal ulceration and SES-CD score of 0-5
Partial clinical response | Month 3, Month 12
  Number of participants with partial clinical response post-injection of 150 or 300 million allogeneic bone marrow derived mesenchymal stem cell product for the treatment of medically refractory Crohn's colitis.
  Partial clinical response is defined as:
  Clinical Healing: >25% reduction of CRP, decrease in CDAI by <100 points
  Radiographic Healing: MR enterography with improvement in inflammation
  Endoscopic healing: Decreased SES-CD by >25% but < 50% or to score of 10-15
Lack of response | Month 3, Month 12
  Number of participants with lack of response post-injection of 150 or 300 million allogeneic bone marrow derived mesenchymal stem cell product for the treatment of medically refractory Crohn's colitis.
  Lack of response is defined as:
  Clinical Healing: No improvement
  Radiographic Healing: MR enterography without resolution of inflammation
  Endoscopic healing: No improvement in SES-CD
Crohn's disease activity index | Month 1 through Month 24
  Crohn's disease activity index will be used to measure quality of life in participants.
  *Remission of Crohn's disease is defined as CDAI below 150. Severe disease is defined as a value of greater than 450.
Inflammatory bowel disease questionnaire | Month 1 through Month 24
  Inflammatory bowel disease questionnaire will be used to measure quality of life in participants.
  *Score ranges from 32 (best health) to 224 (worst health)
EuroQol 5 Dimensions survey | Month 1 through Month 24
  EuroQol 5 Dimensions survey will be used to measure quality of life in participants.
  *Score ranges from 5 (full health) to 25 (worst health).
Inflammatory bowel disease patient reported treatment impact survey | Month 1 through Month 24
  IBD-patient reported treatment impact survey will be used to measure quality of life in participants.
  *Score ranges from 3 (most satisfied) to 15 (least satisfied)
Short Form 36 health survey | Month 1 through Month 24
  Short Form 36 health survey will be used to measure quality of life in participants.
  *Score ranges from 0 (least favorable health state) to 3600 (most favorable health state)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Lightner, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No